CLINICAL TRIAL: NCT03186755
Title: Randomized Controlled Trial Comparing Olopatadine 0.1% Ophthalmic Solution With Hylo-Dual Ophthalmic Preparation in Children With Seasonal Allergic Conjunctivitis
Brief Title: Clinical Evaluation of Hylo-Dual Versus Patanol in Children With Seasonal Allergic Conjunctivitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Marchand, MD (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Michael Marchand, MD, Resident physician in ophthalmology, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-1431
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Conjunctivitis, Allergic; Conjunctivitis, Vernal
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Hyaluronic Acid; Olopatadine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Prospective, Monocentric, Randomized Controlled Trial, Parallel-group, Single-masked for assessors
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hylo-Dual (Experimental): Hyaluronic acid 0.05% & Ectoine 2.0% (Hylo-Dual) 1 drop in both eyes 3 times/day for 8 weeks
  Interventions: Drug: Hyaluronic acid 0.05% & Ectoine 2.0%
- Patanol (Active Comparator): Olopatadine hydrochloride ophthalmic solution 0.1% (Olopatadine) 1 drop in both eyes 2 times/day for 8 weeks
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution 0.1%

INTERVENTIONS:
Drug: Hyaluronic acid 0.05% & Ectoine 2.0% — Treatment of 1 drop three times a day in both eyes for 8 weeks
  Other Names: Hylo-Dual
  Arms: Hylo-Dual
Drug: Olopatadine hydrochloride ophthalmic solution 0.1% — Treatment of 1 drop two times a day in both eyes for 8 weeks
  Other Names: Patanol
  Arms: Patanol

SUMMARY:
This study compares the efficacy of Hylo-Dual (Hyaluronic acid 0.05% & Ectoine 2.0%) and Olopatadine (Olopatadine hydrochloride ophthalmic solution 0.1%) in the control of seasonal allergic conjunctivitis in the pediatric population. Half of participants will receive Hylo-Dual, while the other half will receive Olopatadine treatment for 2 months.

DETAILED DESCRIPTION:
Seasonal allergic conjunctivitis (SAC) is an inflammatory response of the conjunctiva triggered by exposure to seasonal allergens. SAC is the most common form of ocular allergy, with an estimated prevalence of approximately 15 to 20%. The distressing signs (redness, chemosis, eyelid swelling) and symptoms (itching, tearing, redness) of SAC may cause extreme discomfort, with a burden due to the frequency and duration of the disease more than to its seriousness.

Olopatadine hydrochloride ophthalmic solution 0.1% is a topical antiallergic agent that is both an antihistamine with high affinity and selectivity for the histamine H1 receptor and a mast cell stabilizer that inhibits the release of histamine and other proinflammatory mediators from human conjunctival mast cells. The efficacy and tolerability of olopatadine has been demonstrated by several comparative studies in adults and children with seasonal allergic conjunctivitis.

Hylo-Dual eye drops is an approved treatment in Canada for children 6 years and older, containing 0.5mg/ml Sodium Hyaluronate, 20mg/ml Ectoine, a borate buffer and water. Ectoine is a natural substance formed by microorganisms to protect themselves from extreme environments (e.g.: salt lakes or hot geysers). They adapt to these conditions by so-called extremolytes, like ectoine, which are osmoprotective substances stabilizing biological membranes. Ectoine has a strong water-binding capacity, forming a physiologic barrier protecting cell membranes from contact with allergenic substances and against inflammatory responses to environmental stress (such as dehydration, e.g. by hyperosmolar tears, UV radiation or airborne allergens). Additionally, ectoine has a stabilizing effect on the lipid phase of the tear film by increasing its elasticity, which causes it to spread evenly over the eye surface and protects against the excessive evaporation of tears.

To the knowledge of the investigators, no systematic interventional prospective study exists comparing the efficacy of Olopatadine and Hylo-Dual for the treatment of seasonal allergic conjunctivitis in the pediatric population. The research question is to determine if both treatment options are equally effective in this population, therefore providing further clinical pharmacologic data relevant to children.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex and any race aged 6 to 18 years
* History of seasonal allergic conjunctivitis lasting at least 1 allergy season (including patients with rhinoconjunctivitis and atopic dermatitis)
* Current complaint of itching and conjunctival redness in both eyes
* Positive skin reaction to at least one common local grass pollen, including Gramineae, at screening or in the 12 months before the study

Exclusion Criteria:

* Another previous or ongoing ocular disorder
* Presence of significant corneal involvement
* Sensitivity to any component of the study medications
* Use of medication between 1 week before the study and study completion that could confound the interpretation of results (i.e. antihistamines, corticosteroids, nonsteroidal anti-inflammatory drugs, mast cell stabilizers, topical ocular vasoconstrictors)
* Participation in other pharmacologic studies during the month before the study
* Poor baseline visual acuity (not correctable to ≥ 0.6 logMAR in both eyes)
* Autoimmune disease associated with dry eye syndrome (eg, rheumatoid arthritis)
* Inability to discontinue wearing contact lenses during the study
* Inability to discontinue the use of concomitant medication: immunosuppressive drugs, sulfa- or neomycin-containing antibiotics, antibiotics causing allergic reaction

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-06-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Signs of conjunctival erythema | 56 days
  Assessed by an ophthalmologist on slit-lamp examination. 9-point scale consisting of 0.5-unit increments from 0 (normal) to 4 (total involvement). Scale based on the Efron scale.

SECONDARY OUTCOMES:
Signs of conjunctival erythema | 7 days, 14 days, 30 days, 42 days
  Assessed by an ophthalmologist on slit-lamp examination. 9-point scale consisting of 0.5-unit increments from 0 (normal) to 4 (total involvement). Scale based on the Efron scale.
Signs of conjunctival chemosis | 7 days, 14 days, 30 days, 42 days, 56 days
  Assessed by an ophthalmologist on slit-lamp examination. 9-point scale consisting of 0.5-unit increments from 0 (normal) to 4 (total involvement).
Signs of eyelid swelling | 7 days, 14 days, 30 days, 42 days, 56 days
  Assessed by an ophthalmologist on slit-lamp examination. 9-point scale consisting of 0.5-unit increments from 0 (normal) to 4 (total involvement).
Symptoms of itching, self-rated | 7 days, 14 days, 30 days, 42 days, 56 days
  Response to the question, "How often during the last 3 days did your eyes itch enough that you wanted to rub them?" Rated on a 5-point scale.
Symptoms of redness, self-rated | 7 days, 14 days, 30 days, 42 days, 56 days
  Rated by patient or parents on an 11-point scale (VAS - Visual Analog Scale) where 0 = no redness and 10 = the most intense redness imaginable.
Physician's Impression Scale ratings (change scores) | 7 days, 14 days, 30 days, 42 days, 56 days
  Rated on a 6-point scale: 0 = clinical cure, 1 = satisfactory clinical response, 2 = slight clinical improvement, 3 = clinically unchanged, 4 = slightly clinically worse, and 5 = significantly clinically worse.
Listing of adverse effects potentially related to the ophthalmic treatment | 7 days, 14 days, 30 days, 42 days, 56 days
  Based on visual acuity, pupil diameter, intraocular pressure, slit-lamp examination and a dilated fundus examination by an ophthalmologist.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Goodyear, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leonardi A. Emerging drugs for ocular allergy. Expert Opin Emerg Drugs. 2005 Aug;10(3):505-20. doi: 10.1517/14728214.10.3.505. PMID 16083326
- [Background] Leonardi A. Pathophysiology of allergic conjunctivitis. Acta Ophthalmol Scand Suppl. 1999;(228):21-3. doi: 10.1111/j.1600-0420.1999.tb01167.x. No abstract available. PMID 10337426
- [Background] Mortemousque B, Bourcier T, Khairallah M, Messaoud R, Brignole-Baudouin F, Renault D, Rebika H, Bremond-Gignac D; Ketotifen Study Group. Comparison of preservative-free ketotifen fumarate and preserved olopatadine hydrochloride eye drops in the treatment of moderate to severe seasonal allergic conjunctivitis. J Fr Ophtalmol. 2014 Jan;37(1):1-8. doi: 10.1016/j.jfo.2013.02.007. Epub 2013 Dec 31. PMID 24388379
- [Background] Ciprandi G, Turner D, Gross RD. Double-masked, randomized, parallel-group study comparing olopatadine 0.1% ophthalmic solution with cromolyn sodium 2% and levocabastine 0.05% ophthalmic preparations in children with seasonal allergic conjunctivitis. Curr Ther Res Clin Exp. 2004 Mar;65(2):186-99. doi: 10.1016/S0011-393X(04)90032-X. PMID 24764588
- [Background] Bielory L. Update on ocular allergy treatment. Expert Opin Pharmacother. 2002 May;3(5):541-53. doi: 10.1517/14656566.3.5.541. PMID 11996633
- [Background] Bielory L, Lien KW, Bigelsen S. Efficacy and tolerability of newer antihistamines in the treatment of allergic conjunctivitis. Drugs. 2005;65(2):215-28. doi: 10.2165/00003495-200565020-00004. PMID 15631542
- [Background] Katelaris CH, Ciprandi G, Missotten L, Turner FD, Bertin D, Berdeaux G; International Olopatadine Study Group. A comparison of the efficacy and tolerability of olopatadine hydrochloride 0.1% ophthalmic solution and cromolyn sodium 2% ophthalmic solution in seasonal allergic conjunctivitis. Clin Ther. 2002 Oct;24(10):1561-75. doi: 10.1016/s0149-2918(02)80060-1. PMID 12462286
- [Background] McLaurin E, Narvekar A, Gomes P, Adewale A, Torkildsen G. Phase 3 Randomized Double-Masked Study of Efficacy and Safety of Once-Daily 0.77% Olopatadine Hydrochloride Ophthalmic Solution in Subjects With Allergic Conjunctivitis Using the Conjunctival Allergen Challenge Model. Cornea. 2015 Oct;34(10):1245-51. doi: 10.1097/ICO.0000000000000562. PMID 26266427
- [Background] Torkildsen G, Narvekar A, Bergmann M. Efficacy and safety of olopatadine hydrochloride 0.77% in patients with allergic conjunctivitis using a conjunctival allergen-challenge model. Clin Ophthalmol. 2015 Sep 14;9:1703-13. doi: 10.2147/OPTH.S83263. eCollection 2015. PMID 26392751
- [Background] Kam KW, Chen LJ, Wat N, Young AL. Topical Olopatadine in the Treatment of Allergic Conjunctivitis: A Systematic Review and Meta-analysis. Ocul Immunol Inflamm. 2017 Oct;25(5):663-677. doi: 10.3109/09273948.2016.1158282. Epub 2016 May 18. PMID 27192186
- [Background] Bestvater T, Louis P, Galinski EA. Heterologous ectoine production in Escherichia coli: by-passing the metabolic bottle-neck. Saline Syst. 2008 Aug 29;4:12. doi: 10.1186/1746-1448-4-12. PMID 18759971
- [Background] Banciu HL, Sorokin DY, Tourova TP, Galinski EA, Muntyan MS, Kuenen JG, Muyzer G. Influence of salts and pH on growth and activity of a novel facultatively alkaliphilic, extremely salt-tolerant, obligately chemolithoautotrophic sufur-oxidizing Gammaproteobacterium Thioalkalibacter halophilus gen. nov., sp. nov. from South-Western Siberian soda lakes. Extremophiles. 2008 May;12(3):391-404. doi: 10.1007/s00792-008-0142-1. Epub 2008 Feb 29. PMID 18309455
- [Background] Beblo-Vranesevic K, Galinski EA, Rachel R, Huber H, Rettberg P. Influence of osmotic stress on desiccation and irradiation tolerance of (hyper)-thermophilic microorganisms. Arch Microbiol. 2017 Jan;199(1):17-28. doi: 10.1007/s00203-016-1269-6. Epub 2016 Jul 21. PMID 27443666
- [Background] Harishchandra RK, Wulff S, Lentzen G, Neuhaus T, Galla HJ. The effect of compatible solute ectoines on the structural organization of lipid monolayer and bilayer membranes. Biophys Chem. 2010 Aug;150(1-3):37-46. doi: 10.1016/j.bpc.2010.02.007. Epub 2010 Feb 11. PMID 20206435
- [Background] Dwivedi M, Brinkkotter M, Harishchandra RK, Galla HJ. Biophysical investigations of the structure and function of the tear fluid lipid layers and the effect of ectoine. Part B: artificial lipid films. Biochim Biophys Acta. 2014 Oct;1838(10):2716-27. doi: 10.1016/j.bbamem.2014.05.007. Epub 2014 May 20. PMID 24853656
- [Background] Dwivedi M, Backers H, Harishchandra RK, Galla HJ. Biophysical investigations of the structure and function of the tear fluid lipid layer and the effect of ectoine. Part A: natural meibomian lipid films. Biochim Biophys Acta. 2014 Oct;1838(10):2708-15. doi: 10.1016/j.bbamem.2014.05.011. Epub 2014 May 17. PMID 24841755
- [Background] Buenger J, Driller H. Ectoin: an effective natural substance to prevent UVA-induced premature photoaging. Skin Pharmacol Physiol. 2004 Sep-Oct;17(5):232-7. doi: 10.1159/000080216. PMID 15452409
- [Background] DeLuise VP, Peterson WS. The use of topical Healon tears in the management of refractory dry-eye syndrome. Ann Ophthalmol. 1984 Sep;16(9):823-4. PMID 6508097
- [Background] Stuart JC, Linn JG. Dilute sodium hyaluronate (Healon) in the treatment of ocular surface disorders. Ann Ophthalmol. 1985 Mar;17(3):190-2. PMID 3873200
- [Background] Shimmura S, Ono M, Shinozaki K, Toda I, Takamura E, Mashima Y, Tsubota K. Sodium hyaluronate eyedrops in the treatment of dry eyes. Br J Ophthalmol. 1995 Nov;79(11):1007-11. doi: 10.1136/bjo.79.11.1007. PMID 8534643
- [Background] Gill GW, Frost JK, Miller KA. A new formula for a half-oxidized hematoxylin solution that neither overstains nor requires differentiation. Acta Cytol. 1974 Jul-Aug;18(4):300-11. No abstract available. PMID 4135333
- [Background] Papa V, Aragona P, Russo S, Di Bella A, Russo P, Milazzo G. Comparison of hypotonic and isotonic solutions containing sodium hyaluronate on the symptomatic treatment of dry eye patients. Ophthalmologica. 2001 Mar-Apr;215(2):124-7. doi: 10.1159/000050842. PMID 11244343
- [Background] Wysenbeek YS, Loya N, Ben Sira I, Ophir I, Ben Shaul Y. The effect of sodium hyaluronate on the corneal epithelium. An ultrastructural study. Invest Ophthalmol Vis Sci. 1988 Feb;29(2):194-9. PMID 3338879
- [Background] Condon PI, McEwen CG, Wright M, Mackintosh G, Prescott RJ, McDonald C. Double blind, randomised, placebo controlled, crossover, multicentre study to determine the efficacy of a 0.1% (w/v) sodium hyaluronate solution (Fermavisc) in the treatment of dry eye syndrome. Br J Ophthalmol. 1999 Oct;83(10):1121-4. doi: 10.1136/bjo.83.10.1121. PMID 10502570
- [Background] Verin P, Easty DL, Secchi A, Ciprandi G, Partouche P, Nemeth-Wasmer G, Brancato R, Harrisberg CJ, Estivin-Ebrardt C, Coster DJ, Apel AJ, Coroneo MT, Knorr M, Carmichael TR, Kent-Smith BT, Abrantes P, Leonardi A, Cerqueti PM, Modorati G, Martinez M. Clinical evaluation of twice-daily emedastine 0.05% eye drops (Emadine eye drops) versus levocabastine 0.05% eye drops in patients with allergic conjunctivitis. Am J Ophthalmol. 2001 Jun;131(6):691-8. doi: 10.1016/s0002-9394(00)00947-8. PMID 11384563
- [Background] Onguchi T, Dogru M, Okada N, Kato NA, Tanaka M, Takano Y, Fukagawa K, Shimazaki J, Tsubota K, Fujishima H. The impact of the onset time of atopic keratoconjunctivitis on the tear function and ocular surface findings. Am J Ophthalmol. 2006 Mar;141(3):569-71. doi: 10.1016/j.ajo.2005.09.032. PMID 16490512
- [Background] Dogru M, Gunay M, Celik G, Aktas A. Evaluation of the tear film instability in children with allergic diseases. Cutan Ocul Toxicol. 2016 Mar;35(1):49-52. doi: 10.3109/15569527.2015.1010727. Epub 2015 Feb 19. PMID 25694171
- [Background] Nebbioso M, Zicari AM, Celani C, Lollobrigida V, Grenga R, Duse M. Pathogenesis of Vernal Keratoconjunctivitis and Associated Factors. Semin Ophthalmol. 2015;30(5-6):340-4. doi: 10.3109/08820538.2013.874483. Epub 2014 Feb 27. PMID 24571721
- [Background] Gelardi M, Leo ME, Quaranta VN, Iannuzzi L, Tripodi S, Quaranta N, Canonica GW, Passalacqua G. Clinical characteristics associated with conjunctival inflammation in allergic rhinoconjunctivitis. J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):387-91.e1. doi: 10.1016/j.jaip.2015.01.006. Epub 2015 Jan 26. PMID 25634218
- [Background] Bremond-Gignac D, Nischal KK, Mortemousque B, Gajdosova E, Granet DB, Chiambaretta F. Atopic Keratoconjunctivitis in Children: Clinical Features and Diagnosis. Ophthalmology. 2016 Feb;123(2):435-437. doi: 10.1016/j.ophtha.2015.07.012. Epub 2015 Aug 13. No abstract available. PMID 26278858
- [Background] Villani E, Dello Strologo M, Pichi F, Luccarelli SV, De Cilla S, Serafino M, Nucci P. Dry Eye in Vernal Keratoconjunctivitis: A Cross-Sectional Comparative Study. Medicine (Baltimore). 2015 Oct;94(42):e1648. doi: 10.1097/MD.0000000000001648. PMID 26496269
- [Background] Akil H, Celik F, Ulas F, Kara IS. Dry Eye Syndrome and Allergic Conjunctivitis in the Pediatric Population. Middle East Afr J Ophthalmol. 2015 Oct-Dec;22(4):467-71. doi: 10.4103/0974-9233.167814. PMID 26692719
- [Background] Chen L, Pi L, Fang J, Chen X, Ke N, Liu Q. High incidence of dry eye in young children with allergic conjunctivitis in Southwest China. Acta Ophthalmol. 2016 Dec;94(8):e727-e730. doi: 10.1111/aos.13093. Epub 2016 May 26. PMID 27226346
- [Background] Sanchez-Hernandez MC, Montero J, Rondon C, Benitez del Castillo JM, Velazquez E, Herreras JM, Fernandez-Parra B, Merayo-Lloves J, Del Cuvillo A, Vega F, Valero A, Panizo C, Montoro J, Matheu V, Lluch-Bernal M, Gonzalez ML, Gonzalez R, Dordal MT, Davila I, Colas C, Campo P, Anton E, Navarro A; SEAIC 2010 Rhinoconjunctivitis Committee; Spanish Group Ocular Surface-GESOC. Consensus document on allergic conjunctivitis (DECA). J Investig Allergol Clin Immunol. 2015;25(2):94-106. PMID 25997302
- [Background] Vermeulen J, Mercer M. Comparison of the efficacy and tolerability of topical levocabastine and sodium cromoglycate in the treatment of seasonal allergic rhinoconjunctivitis in children. Pediatr Allergy Immunol. 1994 Nov;5(4):209-13. doi: 10.1111/j.1399-3038.1994.tb00241.x. PMID 7894627